CLINICAL TRIAL: NCT01874249
Title: Randomized Clinical Trial to Detect Advanced Fibrosis by Non-invasive Methods in Subjects With Non-alcoholic Fatty Liver Disease
Brief Title: Non Invasive Assessment of Liver Fibrosis in Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Clínica Médica Sur (Other)
Responsible Party: Principal Investigator, Norberto Carlos Chavez Taia, Norberto Carlos Chavez-Tapia, Fundación Clínica Médica Sur
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FAFLD
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Hepatic fibrosis; Steatosis; Noninvasive markers.
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Electronic detailed information (Experimental): Standard of care for patients with diagnosis of fatty liver by ultrasound, plus electronic detailed information about non alcoholic fatty liver disease.
  Interventions: Other: Electronic detailed information
- NAFLD Score (Experimental): Standard of care for patients with diagnosis of fatty liver by ultrasound, plus electronic detailed information about non alcoholic fatty liver disease, plus diagnosis of advanced fibrosis by NAFLD score.
  Interventions: Other: Electronic detailed information; Other: NAFLD Score
- NAFLD Score plus Transient elastography (Experimental): Standard of care for patients with diagnosis of fatty liver by ultrasound, plus electronic detailed information about non alcoholic fatty liver disease, plus diagnosis of advanced fibrosis by NAFLD score and transient elastography.
  Interventions: Other: Electronic detailed information; Other: NAFLD Score; Other: Transient elastography
- Transient elastography (Experimental): Standard of care for patients with diagnosis of fatty liver by ultrasound, plus electronic detailed information about non alcoholic fatty liver disease, plus diagnosis of advanced fibrosis by transient elastography.
  Interventions: Other: Electronic detailed information; Other: Transient elastography
- Standard of care (No Intervention): Standard of care for patients with diagnosis of fatty liver by ultrasound.

INTERVENTIONS:
Other: Electronic detailed information — Electronic detailed information about non alcoholic fatty liver disease.
  Arms: Electronic detailed information; NAFLD Score; NAFLD Score plus Transient elastography; Transient elastography
Other: NAFLD Score — diagnosis of advanced fibrosis by NAFLD score, calculated according to Hepatology 2007;45(4):846-854
  Arms: NAFLD Score; NAFLD Score plus Transient elastography
Other: Transient elastography — Transient elastography values greater than 8 kPa
  Arms: NAFLD Score plus Transient elastography; Transient elastography

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the utility of noninvasive markers for the detection of advanced fibrosis in patients newly diagnosed with Non-alcoholic Fatty Liver Disease (NAFLD) by ultrasound.

The primary objective is to determine the effectiveness of noninvasive markers for detect of advanced fibrosis in patients with diagnosis of fatty liver disease.

The secondary objectives are:

* To determine the increase in health care with the specialist (gastroenterologist or endocrinologist).
* To determine which noninvasive evaluation strategy favors any treatment of fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI ≥ 27 Kg/m2 and any stage of non alcoholic fatty liver, diagnosed by ultrasound.

Exclusion Criteria:

* Patients with other liver disease.
* Patients under treatment with tamoxifen, methotrexate, amiodarone, diltiazem or other drugs able to induce fatty liver.
* Patients with alcohol consumption greater than 140 gr. per week
* Patients who have received blood transfusion before 1990

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2012-07; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Advanced Fibrosis by any diagnostic modality | One year after the diagnosis of steatosis.
  Evidence of advanced fibrosis, diagnosed by transient elastography (greater than 8 kPa), NAFLD Score above 0.675, liver biopsy or any other non-invasive marker of liver fibrosis.

SECONDARY OUTCOMES:
Specialized care | One year after the diagnosis of steatosis.
  Through telephone follow-up, investigate if the patient attends to gastroenterologist or endocrinologist for examination, diagnostic confirmation or any treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Medica Sur Clinic & Foundation, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Chavez-Tapia NC, Barrientos-Gutierrez T, Torres-Ibarra L, Sanchez-Jimenez B, Juarez-Hernandez E, Ramos-Ostos M, Alva-Lopez LF, Uribe M. Incremental levels of diagnostic information incentivize health-seeking in non-alcoholic fatty liver: a randomized clinical trial. Sci Rep. 2022 May 18;12(1):8272. doi: 10.1038/s41598-022-12295-1. PMID 35585153